CLINICAL TRIAL: NCT01434004
Title: A Diet, Physical Activity, and Meditation Intervention in Men With Rising Prostate-specific Antigen
Brief Title: Eating, Activity, and Stress Education
Acronym: EASE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, James hebert, Professor, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: DAMD17-03-1-0139
Record Dates: First submitted 2011-09-07; First posted 2011-09-14 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Prostate Cancer
Keywords: prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lifestyle counseling (Experimental): Diet component: focus on increasing intake of whole grains, soybeans, soybean products, other beans, and vegetables.
  Physical Activity: encourage completion of morning exercise sessions. Mindfulness Stress Reduction: training in mindfulness meditation, including dealing with intensive physical symptoms and difficult emotional situations.
  Interventions: Behavioral: Lifestyle counseling
- Control group (No Intervention): Usual care (watchful waiting).

INTERVENTIONS:
Behavioral: Lifestyle counseling — Diet component: focus on increasing intake of whole grains, soybeans, soybean products, other beans, and vegetables.
  Physical Activity: encourage completion of morning exercise sessions. Mindfulness Stress Reduction: training in mindfulness meditation, including dealing with intensive physical symptoms and difficult emotional situations.
  Arms: Lifestyle counseling

SUMMARY:
The purpose of this study is to determine whether a vegetable-based diet, physical activity program, and stress reduction training will reduce or maintain PSA levels, an indicator of prostate cancer progression, in men who have had their prostate gland removed following a prostate cancer diagnosis.

DETAILED DESCRIPTION:
Following surgery or radiation of a primary early-stage prostate cancer (PrCA), one in three patients will experience an elevation in serum prostate antigen (PSA) within 10 years. For men whose primary treatment was prostatectomy, a PSA rise virtually always signals the spread of PrCA. After such evidence of recurrence, the "standard" treatment is medical or surgical castration. Castration results in reducing the PSA about 85% of the time, but it makes no difference whether such treatment occurs before or after the appearance of clinical symptoms of recurrence. This time interval between the first rise in PSA and symptom appearance may be many years. The most salient fact, however, is that castration does not prolong men's lives and it is not certain whether it even meaningfully delays symptom appearance in men who receive the treatment at the first sign of biochemical recurrence. Castration also has significant side effects including osteoporosis (bone loss), decreased muscle mass, impotence, and urinary incontinence. Because PrCA is usually a disease of older men, many will succumb to other diseases before they ever develop a symptom related to metastatic PrCA. For this large fraction of men, a treatment with deleterious affects on quality of life and no clear overall survival benefit may not be a good choice. The protocol the investigators propose will be performed instead of medical or surgical castration, which is not medically indicated at this point in the course of PrCA. Castration can and will be offered to these men at the first clinical symptom or sign of metastatic cancer, at which time those men will come off this study. It also is important to note that if the intervention results in reductions in PSA then the investigators will offer it to all men who had been randomized to the control condition initially. The investigators will conduct this randomized study in 60 asymptomatic men who have undergone radical prostatectomy (removal of the prostate gland) as their primary therapy of biopsy-confirmed adenocarcinoma of the prostate and subsequently have been found to have rising PSA levels, indicating an early recurrence of the cancer. Half (30) of these men will be randomized to usual care (watchful waiting) and the other half to an intervention consisting of a vegetable-based diet, program of physical activity timed to the natural rhythm of the day (i.e., circadian, or "around the day" - basically to timing of their exercise to improve their sleep cycles), and mindfulness-based stress reduction (consisting of meditation and other stress-reducing techniques). The intervention will continue for three months, followed by monthly booster sessions for 9 months. Data will be collected on compliance with the intervention and other factors that could modify the intervention or confuse our interpretation of its effect. The overall goal of the study will be to see the effect of making these behavioral and attitudinal changes on PSA levels, an indicator of disease progression in these men. The therapies the investigators will study are completely non-toxic and behavioral in nature.

ELIGIBILITY:
Inclusion Criteria:

* have a histologically confirmed diagnosis of adenocarcinoma of the prostate
* have been treated by radical prostatectomy or radiation therapy
* have had no malignancy in the past 5 years (except the primary prostate cancer for which initial treatment was sought and non malignant melanoma of the skin)
* not be taking thyroid medication, antibiotics, diuretics or steroids
* be able to read at a sixth grade level
* speak English as their first language
* be of sound mind, memory, and understanding as evaluated by recruitment staff
* have experienced a rise in serum PSA concentration after achieving a post surgery nadir, after achieving a post radiation nadir, or having had both a radical prostatectomy and subsequent radiotherapy

Exclusion Criteria:

* has received high dose radiotherapy or brachytherapy in place of surgery as a primary treatment
* has received post-operative hormone therapy for prostate cancer
* received treatment of prostate cancer with an LH-RH analog
* has a diagnosis of cardiovascular, pulmonary, or metabolic disease or major symptoms of these diseases, including pain or discomfort in the chest, neck, jaw, arms or other areas that may be due to ischemia; shortness of breath or unusual fatigue at rest or with mild exertion; dizziness; dyspnea while sleeping; ankle edema or intermittent claudication; palpitations, tachycardia, or a known heart murmur
* has experienced a weight loss in excess of five pounds in the previous 3 months
* regularly consumes more than two alcoholic drinks per day
* plans on taking hormone supplements such as melatonin, or fish oil or other; supplements rich in omega-3 fatty acids
* has been diagnosed with Crohn's disease or has active ulcerative colitis
* has been diagnosed with Post Traumatic Stress Disorder (PTSD)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2003-01; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Change in prostate-specific antigen from baseline | baseline, 3 months, 6 months
  PSA is measured at baseline, 3 months and 6 months. Change in PSA is the primary outcome measure.

CONTACTS AND LOCATIONS:
Overall Officials: James R Hebert, Sc.D., Principal Investigator — University of South Carolina
Locations (2):
- United States (2):
  - Palmetto Baptist Medical Center, Columbia, South Carolina
  - Palmetto Richland Memorial Hospital, Columbia, South Carolina